CLINICAL TRIAL: NCT03249272
Title: Microvascular Dysfunction in Nonischemic Cardiomyopathy: Insights From CMR Assessment of Coronary Flow Reserve
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor withdrew funding
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00082447
Record Dates: First submitted 2017-08-08; First posted 2017-08-15 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Hypertrophic Cardiomyopathy; Non-ischemic Dilated Cardiomyopathy; Microvascular Ischaemia of Myocardium
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — regadenoson; Adenosine

STUDY DESIGN:
Intervention Model Description: Participants undergoing cardiovascular magnetic resonance stress testing will be recruited and randomized to receive either regadenoson or adenosine.
Who Masked: Outcomes Assessor
Masking Description: The reader of the CMR scan will be blinded to the stress agent used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hypertrophic cardiomyopathy (Active Comparator)
  Interventions: Drug: Regadenoson; Drug: Adenosine
- Non-ischemic dilated cardiomyopathy (Active Comparator)
  Interventions: Drug: Regadenoson; Drug: Adenosine
- Control (Active Comparator)
  Interventions: Drug: Regadenoson; Drug: Adenosine

INTERVENTIONS:
Drug: Regadenoson — Microvascular disease will be considered present if regional perfusion defects are observed or global perfusion reserve is reduced. For the assessment of microvascular disease, the adenosine and regadenoson groups will be combined, as the medications are considered interchangeable.
Drug: Adenosine — Microvascular disease will be considered present if regional perfusion defects are observed or global perfusion reserve is reduced. For the assessment of microvascular disease, the adenosine and regadenoson groups will be combined, as the medications are considered interchangeable.

SUMMARY:
The aim of this study is to assess microvascular function as determined by a cardiovascular magnetic resonance measurement of whole-heart (global) perfusion reserve. The goal is to determine the prevalence of MVD in two common forms of non-ischemic cardiomyopathy, hypertrophic cardiomyopathy (HCM) and idiopathic dilated cardiomyopathy (IDCM). The hypothesis that an optimized technique will provide robust detection of MVD and that a multifaceted approach will provide new insights into the pathophysiology of MVD, including the influence of myocardial scarring upon the presence and severity of MVD.

DETAILED DESCRIPTION:
Coronary microvascular dysfunction (MVD) has been implicated as an important marker of cardiac risk and has been thought to directly contribute to the pathogenesis of a wide variety of cardiomyopathies. For instance, MVD is believed to cause ischemia (with reduction in coronary flow reserve) in patients with hypertrophic cardiomyopathy (HCM) despite the presence of angiographically normal epicardial coronary arteries. The implication is that MVD in HCM may lead to the ventricular arrhythmias, sudden death, and heart failure. Similarly, patients with idiopathic dilated cardiomyopathy (IDCM) have blunted coronary flow reserve, which appears to be independently associated with poor prognosis.

Several etiologic mechanisms have been proposed to explain the occurrence of MVD, including structural and functional abnormalities1:

1. increased microvascular resistance due to reduced vascular luminal caliber.
2. reduced density of microvessels associated with replacement scarring.
3. inappropriate vasoconstrictor responses.
4. inadequate vasodilator responses.

Unfortunately, these mechanisms are difficult to study in humans since no technique currently allows the direct visualization of the coronary microcirculation in vivo. Thus, MVD has been largely studied using non-invasive imaging techniques, such as positron emission tomography (PET) or single photon emitted computed tomography (SPECT).

Although these methods have provided insight into MVD, much remains unknown. For example, even the prevalence of MVD in patients with various types of cardiomyopathy is unclear, with different studies showing widely different rates.

Cardiovascular magnetic resonance (CMR) is increasingly being used in clinical practice to evaluate cardiac disease. CMR employs a multifaceted imaging approach with separate techniques used to acquire separate sets of raw data, providing information on cardiac morphology, function, regional myocardial ischemia, scarring, and global myocardial perfusion reserve. The advantage of this approach is that image artifacts in one set of data will not affect the quality of the other datasets, and the datasets in combination can be used to distinguish separate pathophysiologies that could confound image interpretation. For example, perfusion defects could be due to ischemia or scar tissue, but since the investigators will obtain both perfusion images and scar images, the investigators will be able to resolve the etiology. Additionally, CMR provides high spatial resolution (over 10-fold higher than PET), and hence partial volume affects will be kept to a minimum and variability in measurements will be reduced.

The aim of this study is to assess microvascular function as determined by a cardiovascular magnetic resonance measurement of whole-heart (global) perfusion reserve. The goal is to determine the prevalence of MVD in two common forms of non-ischemic cardiomyopathy, hypertrophic cardiomyopathy (HCM) and idiopathic dilated cardiomyopathy (IDCM). The hypothesis that an optimized technique will provide robust detection of MVD and that a multifaceted approach will provide new insights into the pathophysiology of MVD, including the influence of myocardial scarring upon the presence and severity of MVD.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years or older

Cardiomyopathy patients

* Patients presenting for CMR with the clinical diagnosis of hypertrophic cardiomyopathy based on left ventricular wall thickness of at least ≥15 mm in the absence of any other cardiac or systemic cause of hypertrophy
* Patients presenting for CMR with the clinical diagnosis of idiopathic dilated cardiomyopathy based upon left ventricular ejection fraction ≤40%, LV end-diastolic diameter ≥55 mm or left ventricular end-systolic diameter ≤45 mm, and the absence of coronary stenoses on angiography.

Control patients

* Patients presenting for CMR without evidence of obstructive coronary artery disease either by coronary angiography or stress testing.

Exclusion Criteria:

* Decompensated heart failure or hemodynamic instability
* Prior coronary revascularization (PCI or CABG) or myocardial infarction (as evidenced by previously elevated CPK-MB or troponin levels)
* Accelerating angina or unstable angina
* Inability to physically tolerate MRI or implanted objects that are MRI incompatible
* Inability to provide written informed consent obtained at time of study enrollment.
* Severe claustrophobia
* Advanced heart block or sinus node dysfunction
* Hypersensitivity or allergic reaction to regadenoson or adenosine
* Hypotension
* Active bronchospasm or history of hospitalization due to bronchospasm
* History of seizures
* Recent cerebrovascular accident
* Use of dipyridamole within the last 5 days
* Contraindication to aminophylline
* Severe renal insufficiency with estimated glomerular filtration rate <30 ml/min/ 1.73 m2
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han Kim, Principal Investigator — Duke University
Locations (1):
- Duke Cardiovascular Magnetic Resonance Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Camici PG, d'Amati G, Rimoldi O. Coronary microvascular dysfunction: mechanisms and functional assessment. Nat Rev Cardiol. 2015 Jan;12(1):48-62. doi: 10.1038/nrcardio.2014.160. Epub 2014 Oct 14. PMID 25311229
- [Background] Klem I, Heitner JF, Shah DJ, Sketch MH Jr, Behar V, Weinsaft J, Cawley P, Parker M, Elliott M, Judd RM, Kim RJ. Improved detection of coronary artery disease by stress perfusion cardiovascular magnetic resonance with the use of delayed enhancement infarction imaging. J Am Coll Cardiol. 2006 Apr 18;47(8):1630-8. doi: 10.1016/j.jacc.2005.10.074. Epub 2006 Mar 27. PMID 16631001
- [Background] Klem I, Greulich S, Heitner JF, Kim H, Vogelsberg H, Kispert EM, Ambati SR, Bruch C, Parker M, Judd RM, Kim RJ, Sechtem U. Value of cardiovascular magnetic resonance stress perfusion testing for the detection of coronary artery disease in women. JACC Cardiovasc Imaging. 2008 Jul;1(4):436-45. doi: 10.1016/j.jcmg.2008.03.010. PMID 19356464
- [Background] Camici PG, Crea F. Coronary microvascular dysfunction. N Engl J Med. 2007 Feb 22;356(8):830-40. doi: 10.1056/NEJMra061889. No abstract available. PMID 17314342
- [Background] Choudhury L, Mahrholdt H, Wagner A, Choi KM, Elliott MD, Klocke FJ, Bonow RO, Judd RM, Kim RJ. Myocardial scarring in asymptomatic or mildly symptomatic patients with hypertrophic cardiomyopathy. J Am Coll Cardiol. 2002 Dec 18;40(12):2156-64. doi: 10.1016/s0735-1097(02)02602-5. PMID 12505229

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to the slow pace of recruitment, the sponsor withdrew funding for the study. Of the expected 75 participants, 31 were recruited. As was pre-specified, the regadenoson and adenosine groups were combined for analysis as these interventions are interchangeable.
Groups:
- Hypertrophic Cardiomyopathy: Microvascular dysfunction (MVD) will be categorized as present based upon the presence of one of the following:
  1. Global perfusion reserve (GPR) < 2.0.
     * Coronary sinus blood flow (CS) with velocity-encoded CMR will be measured during maximal vasodilation and at rest. GPR was calculated as the ratio of stress CS to rest CS blood flow.
  2. The presence of regional perfusion abnormalities on visual assessment of first pass perfusion images.
  For the analysis of the global perfusion ratio, the regadenson and adenosine groups were combined.
  The prevalence will be calculated by dividing the number of hypertrophic cardiomyopathy patients with MVD by the total number of patients with hypertrophic cardiomyopathy.
- Non-ischemic Dilated Cardiomyopathy: Microvascular dysfunction (MVD) will be categorized as present based upon the presence of one of the following:
  1. Global perfusion reserve (GPR) < 2.0.
     * Coronary sinus blood flow (CS) with velocity-encoded CMR will be measured during maximal vasodilation and at rest. GPR was calculated as the ratio of stress CS to rest CS blood flow.
  2. The presence of regional perfusion abnormalities on visual assessment of first pass perfusion images.
  For the analysis of the global perfusion ratio, the regadenson and adenosine groups were combined.
  The prevalence will be calculated by dividing the number of non-ischemic dilated cardiomyopathy patients with MVD by the total number of patients with non-ischemic dilated cardiomyopathy.
- Control: Microvascular dysfunction (MVD) will be categorized as present based upon the presence of one of the following:
  1. Global perfusion reserve (GPR) < 2.0.
     * Coronary sinus blood flow (CS) with velocity-encoded CMR will be measured during maximal vasodilation and at rest. GPR was calculated as the ratio of stress CS to rest CS blood flow.
  2. The presence of regional perfusion abnormalities on visual assessment of first pass perfusion images.
  For the analysis of the global perfusion ratio, the regadenson and adenosine groups were combined.
  The prevalence will be calculated by dividing the number of control patients with MVD by the total number of control patients.
Period: Overall Study
Arm/Group | Hypertrophic Cardiomyopathy | Non-ischemic Dilated Cardiomyopathy | Control
Started | 19 | 6 | 6
Completed | 19 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: As was pre-specified, the regadenoson and adenosine groups were combined for analysis as these interventions are interchangeable.
Groups:
- Hypertrophic Cardiomyopathy: Microvascular dysfunction (MVD) will be categorized as present based upon the presence of one of the following:
  1. Global perfusion reserve (GPR) < 2.0.
     * Coronary sinus blood flow (CS) with velocity-encoded CMR will be measured during maximal vasodilation and at rest. GPR was calculated as the ratio of stress CS to rest CS blood flow.
  2. The presence of regional perfusion abnormalities on visual assessment of first pass perfusion images.
  The prevalence will be calculated by dividing the number of hypertrophic cardiomyopathy patients with MVD by the total number of patients with hypertrophic cardiomyopathy.
- Non-ischemic Dilated Cardiomyopathy: Microvascular dysfunction (MVD) will be categorized as present based upon the presence of one of the following:
  1. Global perfusion reserve (GPR) < 2.0.
     * Coronary sinus blood flow (CS) with velocity-encoded CMR will be measured during maximal vasodilation and at rest. GPR was calculated as the ratio of stress CS to rest CS blood flow.
  2. The presence of regional perfusion abnormalities on visual assessment of first pass perfusion images.
  The prevalence will be calculated by dividing the number of non-ischemic dilated cardiomyopathy patients with MVD by the total number of patients with non-ischemic dilated cardiomyopathy.
- Control Patients: Microvascular dysfunction (MVD) will be categorized as present based upon the presence of one of the following:
  1. Global perfusion reserve (GPR) < 2.0.
     * Coronary sinus blood flow (CS) with velocity-encoded CMR will be measured during maximal vasodilation and at rest. GPR was calculated as the ratio of stress CS to rest CS blood flow.
  2. The presence of regional perfusion abnormalities on visual assessment of first pass perfusion images.
  The prevalence will be calculated by dividing the number of control patients with MVD by the total number of control patients.
- Total: Total of all reporting groups
Arm/Group | Hypertrophic Cardiomyopathy | Non-ischemic Dilated Cardiomyopathy | Control Patients | Total
Number analyzed (Participants) | 19 | 6 | 6 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (17.7) | 60.6 (12.2) | 53.2 (5.7) | 50.3 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 5 | 12
  Male | 14 | 4 | 1 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 4
  White | 16 | 5 | 5 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 5 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Microvascular Dysfunction (MVD) by a CMR Measurement of Whole-heart (Global) Perfusion Reserve Ratio in Patients With Hypertrophic Cardiomyopathy, Non-ischemic Cardiomyopathy, and Controls.
Description: Prevalence of microvascular dysfunction as determined by the CMR measure of global perfusion reserve ratio (GPR) in each these patient groups. MVD was considered present when either GPR was <2.0 or regional stress perfusion abnormalities were present.
  In order to calculate this ratio, coronary sinus flow was measured twice:
  1. prior to the the administration of adenosine/regadenoson
  2. during the administration of adenosine/regadenoson
  GPR is a ratio of coronary sinus flow during the administration adenosine/regadenoson divided by the baseline coronary sinus flow measured prior to the administration.
  Regional perfusion abnormalities will be assessed at the time of adenosine/regadenoson administration.
Time Frame: The prevalence of MVD will be determined based on the findings at the time of the scan on Day 1 of the study.
Population: Due to the slow pace of recruitment, the sponsor withdrew funding for the study. Of the expected 75 participants, 31 were recruited. As was pre-specified, the regadenoson and adenosine groups were combined for analysis as these interventions are interchangeable.
Measure: Number; unit: Percentage of group with MVD
Groups:
- Control: Microvascular dysfunction (MVD) will be categorized as present based upon the presence of one of the following:
  1. Global perfusion reserve (GPR) < 2.0.
     * Coronary sinus blood flow (CS) with velocity-encoded CMR will be measured during maximal vasodilation and at rest. GPR was calculated as the ratio of stress CS to rest CS blood flow.
  2. The presence of regional perfusion abnormalities on visual assessment of first pass perfusion images.
  The prevalence will be calculated by dividing the number of control patients with MVD by the total number of control patients.
Arm/Group | Hypertrophic Cardiomyopathy | Non-ischemic Dilated Cardiomyopathy | Control
Number analyzed (Participants) | 19 | 6 | 5
Percentage of group with MVD | 79 | 33.3 | 20

2. Secondary Outcome: CMR Measurement of Global Perfusion Reserve Ratio
Description: Comparison of the CMR measure of global perfusion reserve ratio (GPR) in each these patient groups.
  In order to calculate this ratio, coronary sinus flow was measured twice:
  1. prior to the the administration of adenosine/regadenoson
  2. during the administration of adenosine/regadenoson
Time Frame: The global perfusion ratio will be calculated from the measurements obtained at the time of the scan on Day 1 of the study.
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: ratio
Groups:
- Hypertrophic Cardiomyopathy; Non-ischemic Dilated Cardiomyopathy; Control: Global perfusion reserve
Arm/Group | Hypertrophic Cardiomyopathy | Non-ischemic Dilated Cardiomyopathy | Control
Number analyzed (Participants) | 19 | 6 | 5
ratio | 2.99 [1.87 to 4.65] | 3.04 [2.64 to 3.61] | 3.83 [2.42 to 4.34]

3. Secondary Outcome: The Association Between Global Perfusion Reserve (GPR) Ratio and Regional Myocardial Scarring.
Description: Relationship between global perfusion reserve ratio and regional myocardial scarring.
Time Frame: Both global perfusion ratio and the presence of regional scarring will be determined/measured from the images obtained during the scan on Day 1 of the study.
Population: As was pre-specified, the regadenoson and adenosine groups were combined for analysis as these interventions are interchangeable. One of the control patients was not able to hold his/her breath, and no image was acquired for stress perfusion myocardial flow. Thus, global perfusion reserve could not be calculated.
Measure: Mean (Standard Deviation); unit: Global perfusion reserve ratio
Groups:
- Hypertrophic Cardiomyopathy - Scarring: Mean value of all patients with Hypertrophic cardiomyopathy with scarring.
- Hypertrophic Cardiomyopathy - Without Scarring: Mean value of all patients with Hypertrophic cardiomyopathy without scarring.
- Non-ischemic Dilated Cardiomyopathy - Scarring: Mean value of all patients with Non-ischemic Dilated cardiomyopathy with scarring.
- Non-ischemic Dilated Cardiomyopathy - Without Scarring: Mean value of all patients with Non-ischemic Dilated cardiomyopathy without scarring.
- Control - Scarring: Mean value of all control patients with scarring.
- Control - Without Scarring: Mean value of all control patients without scarring.
Arm/Group | Hypertrophic Cardiomyopathy - Scarring | Hypertrophic Cardiomyopathy - Without Scarring | Non-ischemic Dilated Cardiomyopathy - Scarring | Non-ischemic Dilated Cardiomyopathy - Without Scarring | Control - Scarring | Control - Without Scarring
Number analyzed (Participants) | 15 | 4 | 6 | 0 | 0 | 5
Global perfusion reserve ratio | 3.19 (1.71) | 5.91 (4.09) | 3.16 (0.65) |  |  | 3.53 (1.26)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during the time of the MR scan.
Groups:
- Hypertrophic Cardiomyopathy - Adenosine; Hypertrophic Cardiomyopathy - Regadenoson; Non-ischemic Dilated Cardiomyopathy - Regadenoson; Control - Regadenoson: Microvascular dysfunction (MVD) will be categorized as present based upon the presence of one of the following:
  1. Global perfusion reserve (GPR) < 2.0.
     * Coronary sinus blood flow (CS) with velocity-encoded CMR will be measured during maximal vasodilation and at rest. GPR was calculated as the ratio of stress CS to rest CS blood flow.
  2. The presence of regional perfusion abnormalities on visual assessment of first pass perfusion images.
  The prevalence will be calculated by dividing the number of hypertrophic cardiomyopathy patients with MVD by the total number of patients with hypertrophic cardiomyopathy.
- Non-ischemic Dilated Cardiomyopathy - Adenosine: Microvascular dysfunction (MVD) will be categorized as present based upon the presence of one of the following:
  1. Global perfusion reserve (GPR) < 2.0.
     * Coronary sinus blood flow (CS) with velocity-encoded CMR will be measured during maximal vasodilation and at rest. GPR was calculated as the ratio of stress CS to rest CS blood flow.
  2. The presence of regional perfusion abnormalities on visual assessment of first pass perfusion images.
  The prevalence will be calculated by dividing the number of non-ischemic dilated cardiomyopathy patients with MVD by the total number of patients with non-ischemic dilated cardiomyopathy.
- Control - Adenosine: Microvascular dysfunction (MVD) will be categorized as present based upon the presence of one of the following:
  1. Global perfusion reserve (GPR) < 2.0.
     * Coronary sinus blood flow (CS) with velocity-encoded CMR will be measured during maximal vasodilation and at rest. GPR was calculated as the ratio of stress CS to rest CS blood flow.
  2. The presence of regional perfusion abnormalities on visual assessment of first pass perfusion images.
  The prevalence will be calculated by dividing the number of control patients with MVD by the total number of control patients.
Arm/Group | Hypertrophic Cardiomyopathy - Adenosine | Hypertrophic Cardiomyopathy - Regadenoson | Non-ischemic Dilated Cardiomyopathy - Adenosine | Non-ischemic Dilated Cardiomyopathy - Regadenoson | Control - Adenosine | Control - Regadenoson
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/2 | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/2 | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/2 | 0/4 | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
Slow recruitment led to the end of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT03249272/Prot_SAP_000.pdf